CLINICAL TRIAL: NCT05843539
Title: Adverse Childhood Experiences, AdaPtatiOn and Breast Cancer
Acronym: CAPONE
Status: Completed | Type: Observational
Sponsor: University of Lorraine (Other)
Collaborators: Ligue contre le cancer, France (Other)
Responsible Party: Principal Investigator, Christine Rotonda, Director of the research pole in Pierre Janet Center, University of Lorraine
Other Study IDs: 2021-A02850-36
Record Dates: First submitted 2023-03-16; First posted 2023-05-06 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Adverse Childhood Experiences; Cancer, Breast; Attachment Styles; Resilience, Psychological; Quality of Life; Epigenesis, Genetic
Keywords: Breast Cancer; ACEs; Quality of Life
MeSH Terms: conditions — Breast Neoplasms | interventions — Biological Products

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — This study also includes a biological ancillary study exploring sub-cellular mechanisms, using high-throughput sequencing to identify gene expression variations that are determinant in terms of vulnerability/protection (cytogenetics and transcriptome).
  The objective of the ancillary study, coupled to the main study, is to show the convergence between self-reported measures related to the presence of ACEs and attachment disorders with assays of chronic stress and epigenetic biomarkers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Genetic: Biological and epigenetic measures — This study also includes an exploratory biological ancillary study that aims to identify the gene expression variations that are determinant in terms of vulnerability/protection (cytogenetic and transcriptome), through the measurement of the level of biological chronic stress and epigenetic methylations of the NR3C1 and FKBP5 genes, in relation to adversity in childhood And to show the convergence between self-reported measures related to the presence of ACEs and attachment disorders with assays of chronic stress and epigenetic biomarkers.

SUMMARY:
Adverse Childhood Experiences (ACEs) have long been linked to mental health problems in adulthood. In the case of cancer, no study has considered that such an anteriority could make patients more vulnerable emotionally, even though the presence of reactionary disorders such as stress, anxiety or depression are characteristic of such a pathology. Activated during periods of stress and therefore during the illness, even the attachment system is mobilized and must be considered to allow more understanding of the illness experience. The attachment style can be seen here as an individual dimension that plays a role in the emotional regulation and resilience of patients. It is also particularly solicited during the remission phase, a complex and singular period of cancer disease that confronts patients with an ambivalence of hope and fear. The fear of recurrence is a concern that the cancer may return or progress in the same organ or in another part of the body. This is a determining factor in the occurrence of anxiety-depressive disorders. Finally, several studies have shown a strong association between depression/anxiety and Cancer-Related Fatigue (CRF) after treatment, especially during the remission phase.

ACEs leave physiological and epigenetic impact that can nowadays be easily evaluated, thus providing additional evidence between adversity, physiological and epigenetic vulnerability and the ability to adapt to life's challenges such as cancer. Life history changes are mediated by changes in cellular mechanisms affecting genome expression. It is currently widely demonstrated that ACEs increases epigenetic modifications.

The interest of this project is therefore to highlight the psychological consequences related to the occurrence of cancer in the developmental history (in terms of adversities) of patients who have completed adjuvant chemotherapy for breast cancer, taking into account the patients' previous attachments, resilience, fear of recurrence and perceived fatigue in order to consider their interactions and their effects on their psychological health and ultimately on their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Have had breast cancer
* Be considered in remission
* Be over 18 years of age
* Literate (able to understand the information and complete the questionnaire independently)
* Agree to participate in the project and sign the informed consent form

Exclusion Criteria:

* Be a person subject to a legal protection measure
* Be a protected adult, under guardianship or curators
* Be undergoing oncological treatment
* Have a lack of autonomy making it impossible to complete the questionnaire online
* Have had or have begun psychotherapeutic treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population studied in this research is a group of adult women who have had breast cancer and are in remission, i.e. whose symptoms and clinical signs visible on medical imaging have diminished or disappeared after treatment for the cancer.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Quality of life of women in remission from breast cancer | Baseline. Through study completion, an average of 1 year.
  The primary outcome was quality of life assessed with the Short Form Survey 12 (SF-12 scale).
  The score ranges from 0 to 100, with a score above 50 indicating average quality of life, 40 to 49 indicating mild disability, 30 to 39 indicating moderate disability, and below 30 indicating severe disability.

SECONDARY OUTCOMES:
Fear of recurrence | Baseline. Through study completion, an average of 1 year.
  The level of fear of cancer recurrence as assessed by the Cancer Recurrence Fear Inventory
Fatigue | Baseline. Through study completion, an average of 1 year.
  Level of fatigue assessed by the Multidimensional Fatigue Inventory (MFI). It is a questionnaire with 20 items on a 5-point likert scale ranging from 1 "strongly disagree" (worth 1 point) to 5 "strongly agree" (worth 5 points). The score is calculated by summing the points on the scale. The higher the score, the more severe the fatigue.
Anxiety and Depression | Baseline. Through study completion, an average of 1 year.
  Level of anxiety and depression assessed using the Hospital Anxiety and Depression Scale (HADS).
  This scale evaluates the level of anxiety in 7 items and the level of depression in 7 items, ranging from 0 to 3. A score greater than or equal to 10 indicates a definite level of anxiety or depression.
Attachment | Baseline. Through study completion, an average of 1 year.
  Attachment relationships were assessed using the Relationship Scales Questionnaire (RSQ).
Adverse Childhood Experiences | Baseline. Through study completion, an average of 1 year.
  The number of adverse childhood and adolescent experiences assessed using the Adverse Childhood Experiences International Questionnaire (ACE-IQ).
  The total number of ACEs to which the participant has been "exposed" is summed to create an ACE score ranging from 0 (no ACEs) to 13. A score of 0 ACEs means a low level of adversity and a score of 13 means a major level of adversity.
Resilience | Baseline. Through study completion, an average of 1 year.
  The level of resilience estimated using the Brief Resilience Scale (BRS). The Brief Resilience Scale is a 6-item questionnaire. Each item is rated on a 5-point Likert scale. Higher scores indicate greater resilience.
RMSSD values | Baseline. Through study completion, an average of 1 year.
  Differences in resting RMSSD (root mean square of successive differences between normal heartbeats) values according to the status with or without ACE, performed via the Caducy (software)

OTHER OUTCOMES:
Stress measurement | Baseline. Through study completion, an average of 1 year.
  Hair cortisol levels via analysis of 100 hairs collected with the root and stored at 4°C
Measurement of epigenetic methylations in relation to childhood adversity | Baseline. Through study completion, an average of 1 year.
  Percentage methylation of genes coding for directed analysis of target regions coding for NR3C1 and FKBP5 genes derived from whole blood, saliva and oral cells assessed using chromatin immunoprecipitation (ChIP) assays

CONTACTS AND LOCATIONS:
Overall Officials: Marion Trousselard, Pr, Principal Investigator — UR 4360 APEMAC, University of Lorraine
Locations (1):
- Ur 4360 Apemac, Metz, Lorraine, France

IPD SHARING:
Plan to Share IPD: No